CLINICAL TRIAL: NCT00799344
Title: Rapid Evaluation of Vessel HEaling After AngiopLasty (REVEAL) Trial: Rationale, Objectives and Design
Brief Title: REVEAL Study: Vessel Healing After Angioplasty
Acronym: REVEAL
Status: Completed | Type: Observational
Sponsor: CeloNova BioSciences, Inc. (Industry)
Responsible Party: Corrado Tamburino, MD, PhD, Ferrarotto Hospital, University of Catania
Other Study IDs: 9 of Nov 24 2008
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stent: Catania Stent
  Interventions: Device: Catania Stent

INTERVENTIONS:
Device: Catania Stent — coronary stent implantation

SUMMARY:
To address early vessel healing and thrombus formation after deployment of three distinct groups of stents

DETAILED DESCRIPTION:
A prospective, randomized study providing new evidences on early vessel healing and thrombus development after stenting with different devices.

ELIGIBILITY:
Inclusion Criteria:

* Lesion length ≤ 20 mm
* Two significant short lesions

Exclusion Criteria:

* Life expectancy < 1 year
* Left ventricular ejection fraction (LVEF) <30%
* Chronic kidney disease

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that have two significant short lesions
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
percentage of "healed stent struts" at 28-32 days | 30 days

SECONDARY OUTCOMES:
Measurement of neointimal growth on stent struts | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Tamburino, MD, Principal Investigator — Ferrarotto Hospital, University of Catania
Locations (1):
- Ferrarotto Hospital, Catania, Sicily, Italy

REFERENCES:
- [Derived] La Manna A, Prati F, Capodanno D, Di Salvo M, Sanfilippo A, Barrano G, Monaco S, Tamburino C. Head-to-head comparison of early vessel healing by optical coherence tomography after implantation of different stents in the same patient. J Cardiovasc Med (Hagerstown). 2011 May;12(5):328-33. doi: 10.2459/JCM.0b013e3283406428. PMID 20962664